CLINICAL TRIAL: NCT03901716
Title: Comparison of Sufentanil, Fentanyl and Remifentanil in Combination With Midazolam During Bronchoscopy Under Conscious Sedation: A Randomized Double-blind Prospective Study
Brief Title: Comparison of Sufentanil, Fentanyl and Remifentanil in Combination With Midazolam During Bronchoscopy Under Conscious Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Clinical Professor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Opioid2019
Record Dates: First submitted 2019-03-30; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Sufentanil; Remifentanil; Fentanyl; Bronchoscopy; Narcotrend; Conscious Sedation
MeSH Terms: interventions — Sufentanil; Fentanyl; Remifentanil; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sufentanil (Experimental): Group S received sufentanil 0.1 mcg/kg and midazolam to achieve moderate levels of sedation as assessed by the Narcotrend (NT; between B1 and C2).
  Interventions: Drug: Sufentanil; Drug: Midazolam
- Fentanyl (Experimental): Group F received fentanyl 1 mcg/kg and midazolam to achieve moderate levels of sedation as assessed by the Narcotrend (NT; between B1 and C2).
  Interventions: Drug: Fentanyl; Drug: Midazolam
- Remifentanil (Experimental): Group R received remifentanil target-controlled infusion with effect-site target concentration of 1ng/ml and midazolam to achieve moderate levels of sedation as assessed by the Narcotrend (NT; between B1 and C2).
  Interventions: Drug: Remifentanil; Drug: Midazolam

INTERVENTIONS:
Drug: Sufentanil — Patients in Group S received sufentanil 0.1 mcg/kg.
  Arms: Sufentanil
Drug: Fentanyl — Patients in Group F received fentanyl 1 mcg/kg.
  Arms: Fentanyl
Drug: Remifentanil — Patients in Group R received remifentanil target-controlled infusion with effect-site target concentration of 1ng/ml.
  Arms: Remifentanil
Drug: Midazolam — Patients in all groups received midazolam to achieve moderate levels of sedation as assessed by the Narcotrend (NT; between B1 and C2).

SUMMARY:
The best opioid for bronchoscopy is still unclear.This randomized double-blind prospective study was conducted on a total of 60 patients who were randomly allocated into 3 groups: Group S received sufentanil 0.1 mcg/kg, Group F received fentanyl 1 mcg/kg and Group R received remifentanil target-controlled infusion with effect-site target concentration of 1ng/ml. Patients in all groups received midazolam to achieve moderate levels of sedation as assessed by the Narcotrend (NT; between B1 and C2). Adverse events, patient tolerance and physician satisfaction were analized.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I-II

Exclusion Criteria:

1. psychological disorders
2. SpO2<90% in ambient air
3. hypersensitivity or allergy to anaesthetic drugs or benzodiazepine
4. severe chronic obstructive pulmonary disease (forced expiratory volume in 1 s ,50% of predicted value, requirement for oxygen therapy)
5. unstable haemodynamic status
6. habitual alcohol consumption
7. asthmatic patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Dosage of midazolam | during the procedure
  Dosage of midazolam applied

SECONDARY OUTCOMES:
severity of cough | during the procedure
  total times of cough
patient's subjective tolerance | 30minutes after bronchoscopy
  the intensity of four key symptoms during bronchoscopy (pain, nausea, breathlessness and cough) and memory using a visual analogic scale (VAS: 1 mm: excellent tolerance, 100 mm very low tolerance)
patient's global tolerance assessed by operator | 30minutes after bronchoscopy
  the global tolerance of patient to the procedure using a visual analogic scale (VAS: 1 mm: excellent tolerance, 100 mm very low tolerance)
rate of oxygen desaturation | during the procedure
  oxygen desaturation (SaO2 decrease<90% for >30 s)

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, Professor, Study Director — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided